CLINICAL TRIAL: NCT02846779
Title: Targeted Adherence Intervention to Reach Glycemic Control With Insulin Therapy for Patients With Diabetes (TARGIT-DM)
Brief Title: Targeted Adherence Intervention to Reach Glycemic Control With Insulin Therapy for Patients With Diabetes
Acronym: TARGIT-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Horizon Blue Cross Blue Shield of New Jersey (Other)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School and Executive Director, Center for Healthcare Delivery Sciences, Department of Medicine, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000648
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Diabetes
Keywords: Insulin persistence; Telepharmacy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ultrasonic Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low intensity (Active Comparator): All participants randomized to this arm will receive quarterly educational mailings and limited telephonic outreach delivered by a pharmacist focused on insulin adherence and glycemic control.
  Interventions: Other: Low intensity
- Moderate intensity (Experimental): Participants will receive all intervention components as in the low-intensity arm but will receive more frequent pharmacist follow-up and the option of enrolling in a text-messaging program. The pharmacist will also provide limited follow-up with the participant's provider. Only 60% of participants randomized will be targeted to receive the intervention based on adherence risk score.
  Interventions: Other: Moderate intensity
- High intensity (Experimental): Participants will receive all intervention components as in the moderate-intensity arm but will receive more frequent pharmacist follow-up. The pharmacist will also provide more follow-up with the participant's provider and/or pharmacist. Only 40% of participants randomized will be targeted to receive the intervention based on adherence risk score and baseline disease control.
  Interventions: Other: High intensity

INTERVENTIONS:
Other: Low intensity — Low intensity telepharmacy outreach
  Arms: Low intensity
Other: Moderate intensity — Moderate intensity telepharmacy outreach
  Arms: Moderate intensity
Other: High intensity — High intensity telepharmacy outreach
  Arms: High intensity

SUMMARY:
The purpose of this study is to evaluate three pharmacist-outreach strategies for improving adherence to insulin among individuals with diabetes. The three approaches are equivalently-priced but vary by degree of targeting and intervention intensity.

DETAILED DESCRIPTION:
In an era of rapidly growing healthcare costs, due to in large part to the increasing burden and complexity of chronic disease management, targeting outreach to patients who are most likely to benefit from them and tailoring interventions to individual patient needs, represent important opportunities to maximize healthcare value. The Targeted Adherence intervention to Reach Glycemic control with Insulin Therapy for patients with Diabetes (TARGIT-DM) trial is a pragmatic, intention-to-treat, randomized-controlled study that will evaluate the impact of three equivalently-priced strategies to improve insulin persistence and glycosylated hemoglobin [HbA1c] control among patients with diabetes on insulin.

The interventions in each of the three study arms will consist of educational mailings and telephonic pharmacist outreach. The pharmacists will assess and address potential barriers to insulin adherence and optimal glycemic control. The three study arms will employ differ both in regards to which patients are targeted and the intensity of the engagement strategy used. The low intensity intervention in arm 1 will be deployed to all subjects randomized to that arm. The moderate and high intensity interventions will be delivered to focused populations within arms 2 and 3, respectively, as defined by poor disease control and/or predicted risk of non-adherence. The interventions provided in the moderate and high intensity arms will also include feedback to the patient's provider, as needed, and potential enrollment in a text messaging program. Patients in these two arms who are not targeted will receive usual care.

The study population for this trial will consist of members enrolled in commercial insurance provided by Horizon Blue Cross Blue Shield of New Jersey. Insurance claims data will be used to apply the inclusion and exclusion criteria. Eligible patients will be randomized into one of three arms, stratified by baseline availability of HbA1c and a valid telephone number.

ELIGIBILITY:
Inclusion Criteria:

* Commercially-insured individuals receiving medical and pharmacy health insurance benefits from Horizon Blue Cross Blue Shield of New Jersey
* At least 3 months of continuous enrollment prior to randomization
* At least 1 prescription for basal insulin, 6 months prior to randomization
* Type 2 diabetes diagnosis

Exclusion Criteria:

* Patients with Medicaid or Medicare as primary insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12-30 (Actual); Study Completion 2018-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Horizon Blue Cross Blue Shield of New Jersey, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauffenburger JC, Lewey J, Jan S, Makanji S, Ferro CA, Krumme AA, Lee J, Ghazinouri R, Haff N, Choudhry NK. Effectiveness of Targeted Insulin-Adherence Interventions for Glycemic Control Using Predictive Analytics Among Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190657. doi: 10.1001/jamanetworkopen.2019.0657. PMID 30874782
- [Derived] Lewey J, Wei W, Lauffenburger JC, Makanji S, Chant A, DiGeronimo J, Nanchanatt G, Jan S, Choudhry NK. Targeted Adherence Intervention to Reach Glycemic Control with Insulin Therapy for patients with Diabetes (TARGIT-Diabetes): rationale and design of a pragmatic randomised clinical trial. BMJ Open. 2017 Oct 30;7(10):e016551. doi: 10.1136/bmjopen-2017-016551. PMID 29084790

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Started | 2000 | 2000 | 2000
Completed | 1861 | 1873 | 1862
Not Completed | 139 | 127 | 138
Not completed — Lost Enrollment | 83 | 82 | 86
Not completed — Less than 31 days of follow-up | 56 | 45 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Intensity | Moderate Intensity | High Intensity | Total
Number analyzed (Participants) | 1861 | 1873 | 1862 | 5596
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.0) | 55.6 (11.3) | 55.9 (10.7) | 55.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 751 | 738 | 763 | 2252
  Male | 1110 | 1135 | 1099 | 3344
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1861 | 1873 | 1862 | 5596
Hemoglobin A1c [Mean (Standard Deviation); unit: % of glycated hemoglobin (A1c)] | 8.5 (1.8) | 8.5 (1.8) | 8.6 (1.8) | 8.5 (1.9)
At least 1 HbA1c value available [Count of Participants; unit: Participants] | 663 | 640 | 642 | 1945
Short or rapid-acting insulin use [Count of Participants; unit: Participants] | 954 | 930 | 965 | 2849
Number of basal insulin claims [Mean (Standard Deviation); unit: Basal insulin claims] | 2.6 (1.9) | 2.6 (1.8) | 2.6 (1.9) | 2.6 (1.9)
Use of adjunct oral hypoglycemic [Count of Participants; unit: Participants] | 1220 | 1242 | 1227 | 3689
Hypoglycemia [Count of Participants; unit: Participants] | 86 | 88 | 87 | 261
Ketoacidosis [Count of Participants; unit: Participants] | 48 | 54 | 41 | 143
Retinopathy [Count of Participants; unit: Participants] | 184 | 156 | 170 | 510
Nephropathy [Count of Participants; unit: Participants] | 46 | 47 | 28 | 121
Neuropathy [Count of Participants; unit: Participants] | 431 | 419 | 412 | 1262
Coronary artery disease [Count of Participants; unit: Participants] | 391 | 405 | 382 | 1178
Hypertension [Count of Participants; unit: Participants] | 1381 | 1409 | 1429 | 4219
Hyperlipidemia [Count of Participants; unit: Participants] | 1278 | 1248 | 1275 | 3801
Congestive heart failure [Count of Participants; unit: Participants] | 129 | 147 | 136 | 412
Stroke/Transient ischemic attack [Count of Participants; unit: Participants] | 95 | 102 | 103 | 300
Obesity [Count of Participants; unit: Participants] | 461 | 472 | 497 | 1430
Asthma/COPD [Count of Participants; unit: Participants] | 254 | 244 | 226 | 724
Cancer [Count of Participants; unit: Participants] | 235 | 221 | 220 | 676
Liver Disease [Count of Participants; unit: Participants] | 130 | 142 | 138 | 410
Chronic Kidney Disease [Count of Participants; unit: Participants] | 1227 | 1222 | 1204 | 3653
Depression [Count of Participants; unit: Participants] | 143 | 135 | 134 | 412
Dementia [Count of Participants; unit: Participants] | 40 | 34 | 36 | 110
Acute Stress [Count of Participants; unit: Participants] | 68 | 62 | 57 | 187
Days hospitalized [Mean (Standard Deviation); unit: Days] | 2.17 (11.1) | 2.2 (10.1) | 2.0 (7.6) | 2.1 (11.0)
Number of Hospitalizations [Mean (Standard Deviation); unit: Hospitalizations] | 0.3 (0.9) | 0.3 (1.3) | 0.3 (0.8) | 0.3 (1.4)
Number of Office visits [Mean (Standard Deviation); unit: Office Visits] | 9.5 (8.0) | 9.3 (7.6) | 9.3 (7.7) | 9.3 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Persistence
Description: Percentage of participants who were non-persistent if they did not refill insulin before a set threshold of time over the entire follow-up period
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Number; unit: Percentage of participants
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 1861 | 1873 | 1862
Percentage of participants | 5.4 | 4.7 | 4.9
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.75 to 1.03]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.77 to 1.06]

2. Secondary Outcome: Change in Glycated Hemoglobin Level (HbA1c)
Description: The percent change in HbA1c level between the latest baseline value to the latest follow up value, among those with at least 1 baseline HbA1c available.
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 663 | 640 | 642
Percent change | -0.06 (1.48) | -0.21 (1.37) | -0.31 (1.48)
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Difference (RD) = -0.15, 95% CI 2-sided [-0.34 to 0.05]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.43 to -0.06]

3. Secondary Outcome: Health Care Spending
Description: Health care spending includes prescription medications, nondrug medical services, and the combination of these two factors over the entire follow-up period
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 1861 | 1873 | 1862
Dollars | 22616 (49250) | 23284 (49094) | 22545 (44448)
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.95 to 1.11]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.92 to 1.06]

4. Secondary Outcome: Number of Physician Office Visits
Description: Number of all-cause physician office visits over the entire follow-up period
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Mean (Standard Deviation); unit: Physician office visits
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 1861 | 1873 | 1862
Physician office visits | 7.66 (7.29) | 7.62 (7.17) | 7.50 (7.27)
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.97 to 1.02]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.96 to 1.00]

5. Secondary Outcome: Number of Emergency Room Visits
Description: Number of all-cause emergency room visits over the entire follow-up period
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Mean (Standard Deviation); unit: ER visits
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 1861 | 1873 | 1862
ER visits | 0.31 (1.00) | 0.43 (4.40) | 0.30 (0.87)
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Ratio (RR) = 1.38, 95% CI 2-sided [1.24 to 1.53]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.85 to 1.07]

6. Secondary Outcome: Number of Hospitalizations
Description: Number of All-cause hospitalizations over the entire follow-up period
Time Frame: From 1 month (30 days) after randomization through 12 months (365 days) after randomization
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
Number analyzed (Participants) | 1861 | 1873 | 1862
Hospitalizations | 0.19 (0.63) | 0.23 (0.72) | 0.21 (0.65)
Statistical Analysis 1: Comparison: Low Intensity vs Moderate Intensity; Test type: Superiority; Risk Ratio (RR) = 1.22, 95% CI 2-sided [1.06 to 1.41]
Statistical Analysis 2: Comparison: Low Intensity vs High Intensity; Test type: Superiority; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.99 to 1.32]

ADVERSE EVENTS:
Time Frame: We did not collect adverse event data (no investigational drug studied). Adverse events were not a pre-specified outcome for the trial. We also did not measure or evaluate mortality.
Description: We did not collect adverse event data (no investigational drug studied). Adverse events were not a pre-specified outcome for the trial. We also did not measure or evaluate mortality.
Arm/Group | Low Intensity | Moderate Intensity | High Intensity
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02846779/Prot_SAP_000.pdf